CLINICAL TRIAL: NCT04437563
Title: Improving Information to Caregivers Via Adaptation and Implementation of the HERMES Intervention the Danish Health Care System
Brief Title: Improving Information to Caregivers Via Adaptation and Implementation of the HERMES Intervention
Acronym: HERMESII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Herlev Gentofte University Hospital, Denmark (Unknown); Rigshospitalet, Denmark (Other); South Jutland Hospital, Denmark (Unknown)
Responsible Party: Principal Investigator, Mogens Groenvold, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R210-A12901
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Cancer; Informal caregivers; Information; Intervention; Stepped wedge cluster randomized controlled trial
MeSH Terms: conditions — Neoplasms | interventions — RBPMS protein, human

STUDY DESIGN:
Intervention Model Description: A stepped wedge cluster randomized controlled trial. All clusters (i.e., participating oncological departments) will start as controls and will change to intervention at various times determined by randomization. In this way, all departments will contribute to control and intervention groups, thus accounting for variation between departments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): ('Standard' care). No intervention offered.
- Intervention (Experimental): ('Standard' care +) The 'Herlev Hospital Empowerment of Relatives through More and Earlier information Supply' (HERMES) intervention.
  Interventions: Behavioral: HERMES

INTERVENTIONS:
Behavioral: HERMES — Via an app, the caregiver answers 14 questions about his/her need for (more) information. The caregiver presents his/her answers (i.e., need for information) to the health care professionals (HCPs), and the HCPs provide the caregiver with the lacking information.
  Arms: Intervention

SUMMARY:
The HERMES intervention was developed in a Danish setting after a comprehensive investigation on caregivers' needs. The intervention consists of: 1) a systematic identification of the caregiver's unmet information needs and 2) a subsequent consultation with a nurse providing the lacking information. The evaluation carried out in a randomized trial at Herlev Hospital showed positive results. It reduced the unmet information needs and improved the caregivers' evaluation of the information from and communication with the health care professionals and the perception of being seen and acknowledged as a caregiver. However, although research projects may show a positive effect, this does not mean that the intervention will be easily implemented in the health care system. Nor does it guarantee that the intervention will show the expected results once implemented in a busy clinical routine.

Therefore, the present project will adapt the HERMES intervention to be implemented in Danish departments of oncology and haematology by (in the first part of the project):

1. Elucidating how the HERMES intervention is best implemented in the clinical setting according to the clinical staff.
2. Elucidating how the HERMES intervention is best implemented in the treatment and follow-up period according to the patients and their caregivers.
3. Developing a technological solution (an app) for the HERMES intervention in which the responses given by the caregivers will form the basis for a subsequent consultation with the health care staff.
4. Revising the HERMES intervention based on the outcomes of a-c.
5. Testing the revised HERMES intervention in a pilot study.

In the second part of the project, the revised HERMES intervention will be tested in a large scale trial with the purpose to:

1. Implement the revised HERMES intervention in the departments of oncology/haematology.
2. Test the effect of the revised HERMES intervention.
3. Evaluate the feasibility of the revised HERMES intervention in a large scale.
4. Elucidate the effectiveness and the feasibility of the intervention and assess possibilities and potential needs for further adaptation in order to secure the future applicability in the Danish Health Care System.

Thus, the overall aim is that by the end of the study, an evidence based and practical implementable method to (continous) use of the HERMES intervention in the Danish health care system is available.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years)
* Primary caregiver (defined as the lay person (partner, family member, friend, etc) most involved in the patient's disease course. The primary caregiver is appointed by the patient)
* Caregiver of an adult cancer patient starting up a treatment course in an oncological department
* Written informed consent to participation

Exclusion Criteria:

* Caregivers not able to read and understand Danish
* Caregivers with no or minimal contact to the oncological department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Quality of information from and communication with health care professionals | Change from baseline (enrollment) to 3 months follow-up
  Measured by the subscale 'Problems with the quality of information from and communication with health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more problems with the quality of information from and communication with health care professionals.

SECONDARY OUTCOMES:
Quality of information from and communication with health care professionals | Change from baseline (enrollment) to 6 months follow-up
  Measured by the subscale 'Problems with the quality of information from and communication with health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more problems with the quality of information from and communication with health care professionals.
Amount of information from health care professionals | Change from baseline (enrollment) to 3 months follow-up
  Measured by (a revised version of) the subscale 'Lack of information from health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of information from health care professionals
Amount of information from health care professionals | Change from baseline (enrollment) to 6 months follow-up
  Measured by (a revised version of) the subscale 'Lack of information from health care professionals' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of information from health care professionals
Attention from health care professionals | Change from baseline (enrollment) to 3 months follow-up
  Measured by the subscale 'Lack of attention from health care professionals on the caregivers' wellbeing' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of attention from health care professionals
Attention from health care professionals | Change from baseline (enrollment) to 6 months follow-up
  Measured by the subscale 'Lack of attention from health care professionals on the caregivers' wellbeing' in the Cancer Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. more lack of attention from health care professionals
Caregiver involvement | Change from baseline (enrollment) to 3 months follow-up
  Measured by item 12 in the Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item score range: 0-100. A higher score represents a worse outcome, i.e. more caregiver dissatisfaction with involvement
Caregiver involvement | Change from baseline (enrollment) to 6 months follow-up
  Measured by item 12 in the Caregiving Tasks, Consequences and Needs Questionnaire (CaTCoN). Item score range: 0-100. A higher score represents a worse outcome, i.e. more caregiver dissatisfaction with involvement
Emotional functioning | Change from baseline (enrollment) to 3 months follow-up
  Measured by the European Organisation for Research and Treatment of Cancer (EORTC) Emotional Functioning 10 scale (EORTC EF10). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. worse emotional functioning
Emotional functioning | Change from baseline (enrollment) to 6 months follow-up
  Measured by the EORTC Emotional Functioning 10 scale (EORTC EF10). Subscale score range: 0-100. A higher score represents a worse outcome, i.e. worse emotional functioning
Positive emotional functioning | Change from baseline (enrollment) to 3 months follow-up
  Measured by a scale of five positively formulated items concerning emotional functioning which were excluded from the EORTC Computerized Adaptive Test (CAT) emotional functioning bank during the development of the item bank. Subscale score range: 0-100. A higher score represents a better outcome, i.e. more positive emotional functioning
Positive emotional functioning | Change from baseline (enrollment) to 6 months follow-up
  Measured by a scale of five positively formulated items concerning emotional functioning which were excluded from the EORTC Computerized Adaptive Test (CAT) emotional functioning bank during the development of the item bank. Subscale score range: 0-100. A higher score represents a better outcome, i.e. more positive emotional functioning

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Groenvold, PhD DMSc, Principal Investigator — Bispebjerg and Frederiksberg Hospital, University of Copenhagen
Locations (8):
- Denmark (8):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Hospitalsenheden Vest, Herning
  - Naestved Sygehus, Næstved
  - Roskilde Universitetshospital, Roskilde
  - Sygehus Soenderjylland, Sønderborg
  - Vejle Sygehus, Vejle